CLINICAL TRIAL: NCT01723384
Title: Intermittent Naltrexone Among Polysubstance Users
Acronym: Project iN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Glenn-Milo Santos, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-09809; R36DA035109-01 (NIH)
Record Dates: First submitted 2012-11-02; First posted 2012-11-07 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Methamphetamine; Alcohol
Keywords: methamphetamine; alcohol; HIV; sexual behavior
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Active Comparator): Intermittent oral naltrexone to be taken on an as-needed basis for 8 weeks.
  Interventions: Drug: Intermittent Oral Naltrexone
- Placebo (Placebo Comparator): Intermittent oral placebo to be taken on an as-needed basis for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intermittent Oral Naltrexone
  Arms: Naltrexone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Naltrexone, a µ-opioid receptor antagonist, is a promising agent for methamphetamine-using and binge-drinking men who have sex with men (MSM). Naltrexone has shown efficacy in reducing relapse to amphetamines and is FDA-approved for alcohol dependence. Oral naltrexone is inexpensive and has few toxicities but the standard daily regimen for naltrexone is problematic as patients forget to take the medication. Given the challenges in daily dosing, alternate regimen schedules have been proposed to increase efficacy and expand the population that may benefit from this pharmacologic agent. One approach is intermittent targeted administration of naltrexone, whereby individuals take the medication as-needed in anticipation of substance use or during periods of craving. Administration of naltrexone prior to exposure to amphetamines significantly attenuates craving and targeted naltrexone has shown efficacy in reducing heavy alcohol use. However, there have been no studies assessing intermittent targeted dosing of naltrexone among methamphetamine-using and binge-drinking MSM. Polysubstance use patterns are common among MSM, and studies among those who abuse more than one substance are urgently needed. The aims of this study are to determine whether targeted dosing of naltrexone is feasible, tolerable and acceptable among non-dependent methamphetamine-using and binge-drinking MSM.

ELIGIBILITY:
Inclusion Criteria:

1. male gender or transgender male-to-female
2. self-reported anal sex with men in the prior six months while under the influence of meth and/or alcohol
3. self-reported meth use at least bi-weekly in the prior three months
4. at least weekly binge drinking (five or more drinks on a single drinking session) in the prior three months

4) interested in reducing meth use and/or binge drinking 5) HIV-negative by rapid test or medical record of HIV infection 6) no current acute illnesses requiring prolonged medical care 7) no chronic illnesses that are likely to progress clinically during trial participation 8) able and willing to provide informed consent and adhere to visit schedule 9) age 18-70 years 10) baseline complete blood count (CBC), total protein, albumin, glucose, alkaline phosphatase, creatinine, blood urea nitrogen (BUN), and electrolytes without clinically significant abnormalities as determined by study clinician in conjunction with symptoms, physical exam, and medical history

Exclusion Criteria:

1. any psychiatric (e.g., depression with suicidal ideation) or medical condition that would preclude safe participation in the protocol
2. known allergy or previous adverse reaction to naltrexone
3. current use of or dependence on any opioids or a known medical condition which currently requires or may likely require opioid analgesics
4. opioid-positive urine test at enrollment
5. current cluster of differentiation 4 (CD4) count < 200 cells/mm3
6. moderate or severe liver disease (aspartate aminotransferase, alanine aminotransferase, or total bilirubin > 3 times upper limit of normal)
7. impaired renal function (creatinine clearance < 60 ml/min)
8. currently participating in another research study
9. meth or alcohol dependence as determined by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (SCID) criteria
10. any condition that, in the principal investigator and/or study clinician's judgment interferes with safe participation or adherence to study procedures.
11. unwillingness to provide minimum locator for information
12. not having a cellular phone that can send or receive a text message
13. plans to leave the Bay Area during study follow-up
14. not comfortable speaking and reading English, enough to participate in a program in English

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn-Milo Santos, PhD, Principal Investigator — University of California, San Francisco; Jason Euren, MA, Study Director — San Francisco Department of Public Health
Locations (1):
- San Francisco Department of Public Health, Substance Use Research Unit, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone: Intermittent oral naltrexone to be taken on an as-needed basis for 8 weeks.
  Intermittent Oral Naltrexone
- Placebo: Intermittent oral placebo to be taken on an as-needed basis for 8 weeks
  Placebo
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (10) | 42.3 (10) | 43 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Retaining Participants in Trial
Description: Proportion of persons retained by study arm.
Time Frame: proportions eligible and enrolled assessed on ongoing basis throughout the study, proportion of visits completed assessed bi-weekly for each participant; overall retention assessed over 2 month follow-up for each participant
Measure: Number; unit: percentage that completed study
Groups:
- Naltrexone: Naltrexone
- Placebo: Placebo
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 15 | 15
percentage that completed study | 100 | 86.7

2. Primary Outcome: Acceptability to Taking Medication
Description: Mean number of pills taken weekly, as determined by recorded openings from an electronic monitoring device for study medication pill dispensers
Time Frame: 2 month follow-up
Measure: Mean (Standard Deviation); unit: number of wisepill openings by week
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 15 | 15
number of wisepill openings by week | 2.2 (1) | 1.9 (1)

3. Primary Outcome: Tolerability to Study Drug, as Measured by Adverse Events
Description: Frequency of Adverse Events, by arm
Time Frame: 2 months
Measure: Number; unit: Count
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 15 | 15
Count
  Nausea | 4 | 2
  Headaches | 2 | 1
  Upper respiratory tract infection | 2 | 4

ADVERSE EVENTS:
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 8/15 | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=15) | Placebo (N=15)
Nausea (General disorders) | 4 (4) | 2 (2)
Headaches (General disorders) | 2 (2) | 1 (1)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No